CLINICAL TRIAL: NCT00492024
Title: Prospective, Multicenter, Randomized, Double-Blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Moxifloxacin 400 mg QD for 5 Days Versus Placebo in the Treatment of Acute Bacterial Sinusitis
Brief Title: BAY12-8039: 5 Days for Sinusitis vs Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11566
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2009-12-02 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Sinusitis
Keywords: Respiratory Tract Infection; Bacterial Sinusitis
MeSH Terms: conditions — Sinusitis; Respiratory Tract Infections | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin 400 mg (Experimental): Moxifloxacin 400mg once daily for 5 days
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)
- Placebo (Placebo Comparator): Matching placebo for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Moxifloxacin - 400 mg once a day for 5 days
  Arms: Moxifloxacin 400 mg
Drug: Placebo — Placebo - 380 mg Microcrystalline Cellulose
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of Avelox in a 5 day treatment of adult patients with acute bacterial sinusitis and to measure the amount of time it takes for symptom relief. Avelox is currently not approved for the 5 day treatment of acute bacterial sinusitis, therefore in this study Avelox is considered an investigational drug. In this study Avelox will be compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria at the time of enrollment:

* Age >/= 18 years
* Clinical diagnosis of acute bacterial sinusitis with signs and symptoms present for = 7 days but < 28 days as defined by A), radiographic, and B) clinical criteria, as follows:

  * Radiographic Criteria: The presence of one or more of the following on a radiographic paranasal sinus film (Waters' view): - Evidence of air-fluid levels - Opacification
  * Clinical Criteria: The presence of two major symptoms, or the presence of at least one major and one minor symptom as defined in the list below:

    * Major symptoms: - Purulent anterior or posterior nasal discharge - Unilateral facial pain or malar tenderness
    * Minor symptoms: - Frontal headache - Fever (oral = 38.0°C/100.4°F, tympanic = 38.5°C/101.2°F, axillary = 37.5°C/99.5°F) - Culture material obtained by sinus puncture; the aspirated specimen sent for Gram stain, quantitative culture and susceptibility testing prior to initiation of antimicrobial therapy

Exclusion Criteria:

Subjects with one or more of the following criteria will not be eligible for this study:

* History of chronic sinusitis defined as greater than four weeks of continuous symptoms (subjects with recurrent acute sinusitis will be included)
* History of sinus surgery (antral sinus puncture is not considered as a surgery)
* Any symptoms that suggest the subject's current illness is allergic rhinitis (e.g. repetitive sneezing, itchy nose or eyes, provocation by an allergen) and not acute bacterial sinusitis
* Known bacteremia, meningitis or infection infiltrating the tissues neighboring the sinuses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2005-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (48):
- United States (48):
  - Birmingham, Alabama
  - Northport, Alabama
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Fresno, California
  - Garden Grove, California
  - Orange, California
  - Roseville, California
  - San Diego, California
  - San Luis Obispo, California
  - Colorado Springs, Colorado
  - Bridgeport, Connecticut
  - Dunnellon, Florida
  - Hialeah, Florida
  - North Miami Beach, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - Atlanta, Georgia
  - Warner Robbins, Georgia
  - Warner Robins, Georgia
  - Louisville, Kentucky
  - Detroit, Michigan
  - Livonia, Michigan
  - Portage, Michigan
  - Butte, Montana
  - Elizabeth, New Jersey
  - Lawrenceville, New Jersey
  - Somerville, New Jersey
  - Rochester, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Eugene, Oregon
  - Levittown, Pennsylvania
  - Norristown, Pennsylvania
  - Palmyra, Pennsylvania
  - Clarksville, Tennessee
  - Austin, Texas
  - College Station, Texas
  - El Paso, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Tappahannock, Virginia
  - Bellingham, Washington
  - Greenfield, Wisconsin

REFERENCES:
- [Result] Hadley JA, Mosges R, Desrosiers M, Haverstock D, van Veenhuyzen D, Herman-Gnjidic Z. Moxifloxacin five-day therapy versus placebo in acute bacterial rhinosinusitis. Laryngoscope. 2010 May;120(5):1057-62. doi: 10.1002/lary.20878. PMID 20422704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 37 investigative centers in the United States from January 2005 to March 2008.
Pre-assignment Details: Modified Intent-to-Treat (MITT): Subjects who received at least 1 dose of study drug with a baseline sinus culture positive for at least 1 of 5 common bacteria that cause sinusitis (73 moxifloxacin [M], 45 placebo [P]). Per protocol (PP): Subjects with a positive baseline culture (as above) meeting a long list of additional criteria (62 M, 42 P).
Period: Treatment
Arm/Group | Moxifloxacin 400 mg | Placebo
Started | 251 | 123
Completed | 222 | 101
Not Completed | 29 | 22
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 21 | 20
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Period: Follow up
Arm/Group | Moxifloxacin 400 mg | Placebo
Started | 222 | 101
Completed | 221 | 99
Not Completed | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin 400 mg | Placebo | Total
Number analyzed (Participants) | 251 | 123 | 374
Age Continuous [Mean (Standard Deviation); unit: years] | 40.1 (13.8) | 40.3 (13.0) | 40.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 80 | 245
  Male | 86 | 43 | 129
Causative Organisms Isolated from Pretreatment Specimens at Study Entry [Number; unit: participants] — Causative organisms identified by pre-therapy sinus puncture (more than one organism was identified for some patients)
  participants
    Streptococcus pneumoniae | 32 | 13 | 45
    Moraxella catarrhalis | 7 | 12 | 19
    Haemophilus influenzae | 28 | 15 | 43
    Streptococcus pyogenes | 2 | 2 | 4
    Staphylococcus aureus | 11 | 5 | 16
    Non causative pathogene | 66 | 32 | 98
    No pathogene growth | 109 | 45 | 154
Location of infection [Number; unit: participants] — Location of sinus infection, left, right, or bilateral
  participants
    Left | 82 | 37 | 119
    Right | 94 | 46 | 140
    Bilateral | 75 | 40 | 115
Severity of infection [Number; unit: participants] — Severity of infection as asessed by the investigator
  participants
    Moderate | 153 | 72 | 225
    Severe | 90 | 49 | 139
    Mild | 8 | 2 | 10
Duration of infection [Mean (Standard Deviation); unit: days] — Subgroup analyses were performed on subjects with differing durations of infection of 7 to 14 days, 15 to 21 days, and 22 to 27 days.
  days | 13.2 (5.4) | 12.7 (4.7) | 13.0 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Clinical Cure (Modified Intent-to-Treat (MITT))
Description: The primary efficacy variable was clinical response (CR) at the TOC visit, and was rated as improvement, complete resolution, failure, or indeterminate. Clinical cure, ie, success, was defined as complete resolution or improvement in the signs and symptoms such that no further therapy (antimicrobial, steroid, or irrigation) was required.
Time Frame: At 'Test-of-Cure' (TOC), Day 1-5 after end of treatment
Population: The modified intent-to-treat (MITT) population was the primary analysis population. This population includes all subjects treated with at least one dose of study medication, and who have at least one pre-treatment causative organism.
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 73 | 45
Percentage of subjects
  Success (Clinical Cure) | 78.1 | 66.7
  Failure | 19.2 | 33.3
  Indeterminate | 2.7 | 0
  Complete resolution | 12.3 | 11.1
  Improvement | 65.8 | 55.6
Statistical Analysis 1: Comparison: Moxifloxacin 400 mg vs Placebo; Null hypothesis is that the success rate for moxifloxacin = the success rate for placebo; Test type: Superiority or Other; p = 0.189, Cochran-Mantel-Haenszel — P-value is adjusted for study center; p-value applies to percentage of subjects with success (clinical cure); Adjusted for study center

2. Secondary Outcome: Treatment Day When Patients Reached Symptom Improvement as Measured by Patient Reported Data, Using Last Observation Carried Forward (LOCF) Approach
Description: The Sino-Nasal Outcome Test (SNOT-16) was used to assess subject-reported time to symptom improvement. Improvement was defined as a decrease of at least 14 units on the test. This difference is the smallest difference that has been identified as beneficial to subjects.
Time Frame: Daily until 'Test-Of-Cure' (Day 1-5 after end of treatment)
Population: The MITT population was the primary analysis population. This population includes all subjects treated with at least one dose of study medication, and who have at least one pre-treatment causative organism.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 73 | 45
participants
  Day 2 | 14 | 7
  Day 3 | 26 | 10
  Day 4 | 31 | 13
  Day 5 | 39 | 16
  Test-Of-Cure | 43 | 19

3. Secondary Outcome: Treatment Day When Patients Returned to Normal Activities as Measured by Patient Reported Data, Using LOCF Approach
Description: The Activity Impairment Assessment (AIA) questionnaire was used to assess activity impairment at baseline and time to return to normal activities. The AIA was administered prior to first dose, every 24 hours during treatment, and at the TOC visit. Improvement in the AIA total score was defined as a decrease of at least 3 units.
Time Frame: Daily until 'Test-Of-Cure' (Day 1-5 after end of treatment)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 73 | 45
participants
  Day 2 | 22 | 15
  Day 3 | 31 | 17
  Day 4 | 35 | 17
  Day 5 | 37 | 19
  Test-Of-Cure | 42 | 22

4. Secondary Outcome: Percentage of Subjects With Clinical Improvement During Therapy
Description: A secondary efficacy variable was clinical response (CR) at the During Therapy visit at day 3 or 4 of treatment. CR was rated as improvement, cure, failure, or indeterminate. Clinical evaluation was based on the presence and severity (mild, moderate, or severe) of several signs and symptoms of acute sinusitis.
Time Frame: Day 3 of treatment
Population: The MITT population was the primary analysis population. This population includes all subjects treated with at least one dose of study medication, and who have at least one pre-treatment causative organism. Missing responses at during therapy visit in most cases was due to early clinical failure.
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 73 | 45
Percentage of subjects
  Improvement | 84.9 | 73.3
  Indeterminate | 4.1 | 4.4
  Missing | 11.0 | 22.2

5. Secondary Outcome: Percentage of Subjects With Continued Clinical Cure During Long-Term Follow-Up
Description: A secondary efficacy variable was clinical response (CR) at the Follow-up visit 17-21 days following the start of treatment. CR was rated as continued cure, failure/relapse, or indeterminate. Clinical evaluation was based on the presence and severity (mild, moderate, or severe) of several signs and symptoms of acute sinusitis.
Time Frame: Day 12 to 26 after end of treatment
Population: as for outcome 2
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 73 | 45
Percentage of subjects
  Combined Clinical Cure | 73.9 | 57.7
  Clinical Failure / Relapse | 21.9 | 40.0
  Missing | 4.1 | 2.2

6. Other Pre Specified Outcome: Percentage of Subjects With Clinical Cure (Per Protocol Population (PP))
Description: as for outcome 1
Time Frame: At 'Test-of-Cure', Day 1-5 after end of treatment
Population: This analysis population was per protocol population, which included all subjects with at least one pre-treatment causative organism, and who had no major deviations from the protocol procedures.
Measure: Number; unit: Percentage of subjects
Arm/Group | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 62 | 42
Percentage of subjects
  Success | 82.3 | 66.7
  Failure | 17.7 | 33.3
  Indeterminate | 0 | 0
  Complete resolution | 11.3 | 9.5
  Improvement | 71.0 | 57.1
Statistical Analysis 1: Comparison: Moxifloxacin 400 mg vs Placebo; Null hypothesis is that the success rate for moxifloxacin = the success rate for placebo; Test type: Superiority or Other; p = 0.075, Cochran-Mantel-Haenszel — p-value adjusted for study center; p-value applies to percentage of subjects with success (clinical cure); adjusted for study center

ADVERSE EVENTS:
Arm/Group | Moxifloxacin 400 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/251 | 1/123
Other Adverse Events (participants affected / at risk) | 49/251 | 23/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moxifloxacin 400 mg (N=251) | Placebo (N=123)
Pneumonia (Infections and infestations) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moxifloxacin 400 mg (N=251) | Placebo (N=123)
Nausea (Gastrointestinal disorders) | 11 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 3 | 3
Procedural Pain (Injury, poisoning and procedural complications) | 6 | 6
Headache (Nervous system disorders) | 11 | 4
Dizziness (Nervous system disorders) | 9 | 1
Sinus headache (Nervous system disorders) | 6 | 2
Insomnia (Psychiatric disorders) | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2

LIMITATIONS AND CAVEATS:
Confounding factors include concomitant medication for symptomatic relief not standardised, TOC visit occured earlier than for other sinusitis studies, response on placebo underestimated and short-term relief provided by the sinus tap.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days